CLINICAL TRIAL: NCT01032252
Title: Prevention of Falls in Community-dwelling Older Adults by a Standardized Assessment of Fall Risks in the General Practitioner Setting and Through Implementation of a Network for Effective Individual Reduction on Fall Risks.
Brief Title: Prevention of Falls in General Practitioner for Community-dwelling Older Adults [PreFalls]
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FAU061209TUM; FAU061209TUM (Other Grant/Funding Number: Bavarian State Ministry of the Environment and Public Health)
Record Dates: First submitted 2009-12-12; First posted 2009-12-15 (Estimated); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Accidental Falls/Prevention & Control; Risk Assessment; General Practitioner Education; Humans; Multicenter Study; Randomized Controlled Trial
Keywords: fall prevention; general practitioners setting; implementation; network; community dwelling older adults; exercise intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- observational (No Intervention): Control group: followed by monthly falls calenders and four testing periods
- Exercise group (Experimental): 16 week intervention, and followed by monthly fall calenders as well as 4 testing periods
  Interventions: Other: Exercise intervention

INTERVENTIONS:
Other: Exercise intervention — 16 week exercise once a week of 60 minutes intervention by trained fall prevention instructors and a home program.
  Intervention includes strength/power training, balance/gait training, behavioral aspects and perceptual and functional training.
  Arms: Exercise group

SUMMARY:
The primary aim of this two-year project for falls prevention is to reduce number of falls and fall incidence in community-dwelling people of 65 years and older in the setting of general practitioners. In addition a reduction of fall-related injuries, reduction of fall-related risk factors and preservation of Quality of Life is to be achieved.

A second goal of this study is the implementation of standardized assessment for fall risk factors as well as building up a network between instructors for fall prevention exercise and general practitioners.

DETAILED DESCRIPTION:
Health related consequences of falls are underestimated. In comparison to different health related risk factors like hypertension etc. falls and their risks are being underestimated by many physicians. Regardless of the high relevance of falls for the elderly as well as the Health Care System, risk of falling is only rarely being assessed. The reasons for this are manifold. Insufficient assessment of risk of falling are one of the reasons. Many registered doctors with their own practice do not use a standardized assessment of risk of falling that is quick and effective. Additionally, patients rarely report occurred falls to their physicians because they don't know the implications or are afraid of subsequently losing their independence.

Physicians already assessing their senior patients' risk of falling lack the possibility to assign them to according ambulatory interventions since these scarcely exist in Bavaria. Chances for improvement are: standardized assessment of risk of falling needed to uncover senior patients' risk of falling quickly, reliably and efficiently at their family physician's. At the same time area-wide programs to effectively reduce falls by targeting individual behavior as well as general conditions must be provided to maintain the independence of individual senior citizens.

ELIGIBILITY:
Inclusion Criteria:

* Target group are community-dwelling senior citizens aged 65 years or above with an increased risk of falling.
* Increased risk of falling are seen by:

  * history of falls
  * fear of falling
  * chair rise > 10 sec./TUG > 10 sec./ subjective & objective balance deficits

Exclusion Criteria:

* Elderly people not living independently or suffering from physical or mental restrictions that do not allow the participation in an exercise program or the assessment of risk of falling

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 378 (Actual)
Dates: Start 2009-04; Primary Completion 2011-09 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Primary outcomes are number of falls and falls rates as well as number and incidence of injurious falls measured by monthly fall calendars | 24 months

SECONDARY OUTCOMES:
Secondary endpoints are a reduction in fear of falling, a reduction in risk of falling in the physical dimensions e.g. strength, balance and function, the preservation of quality of life and the preservation or increase in physical activity. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Monika Siegrist, PhD, Principal Investigator — Department of Medicine, Division of Prevention and Sports Medicine TU Munich; Ellen Freiberger, PhD, Principal Investigator — Department of Sport Science, University of Erlangen-Nürnberg
Locations (1):
- Department of Medicine, Division of Prevention and Sports Medicine TU Munich, Munich, Germany

REFERENCES:
- [Background] Blank WA, Freiberger E, Siegrist M, Landendoerfer P, Linde K, Schuster T, Pfeifer K, Schneider A, Halle M. An interdisciplinary intervention to prevent falls in community-dwelling elderly persons: protocol of a cluster-randomized trial [PreFalls]. BMC Geriatr. 2011 Feb 17;11:7. doi: 10.1186/1471-2318-11-7. PMID 21329525